CLINICAL TRIAL: NCT02016625
Title: Investigation of Potential Drug-drug Interactions Between Faldaprevir and Immunosuppressants (Cyclosporine and Tacrolimus) in Healthy Male and Female Subjects (Open-label, Fixed-sequence Trial)
Brief Title: Investigation of Potential Drug-drug Interactions Between Faldaprevir and the Immunosuppressant Drugs Cyclosporine or Tacrolimus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1241.61; 2013-003435-30 (EudraCT Number: EudraCT)
Record Dates: First submitted 2013-12-16; First posted 2013-12-20 (Estimated); Results first posted 2016-04-18 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-04

CONDITIONS: Healthy
MeSH Terms: interventions — faldaprevir; Cyclosporine; Tacrolimus

ARMS (2):
- 1 Cyclosporine + Faldaprevir (Experimental)
  Interventions: Drug: Faldaprevir; Drug: Cyclosporine
- 2 Tacrolimus + Faldaprevir (Experimental)
  Interventions: Drug: Faldaprevir; Drug: Tacrolimus

INTERVENTIONS:
Drug: Faldaprevir
  Arms: 1 Cyclosporine + Faldaprevir
Drug: Faldaprevir
  Arms: 2 Tacrolimus + Faldaprevir
Drug: Cyclosporine
  Arms: 1 Cyclosporine + Faldaprevir
Drug: Tacrolimus
  Arms: 2 Tacrolimus + Faldaprevir

SUMMARY:
The primary objective of this trial is to investigate the effect of multiple-dose faldaprevir (FDV) on the single-dose pharmacokinetics of cyclosporine or tacrolimus

ELIGIBILITY:
Inclusion criteria:

* Healthy males or females subjects
* Age 18 to 50 years (incl.)
* Body mass index (BMI) 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study

Exclusion criteria:

* Any finding in the medical examination (including blood pressure, pulse rate or ECG) deviating from normal and judged clinically relevant by the investigator.
* Systolic blood pressure (BP) less than 100 mmHg and more than 140 mmHg.
* Diastolic BP less than 60 mmHg and more than 90 mmHg.
* Pulse rate (PR) less than 50 bpm and more than 90 bpm.
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged clinically relevant by the investigator
* Positive QuantiFERON-TB Gold In-Tube

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2013-12; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1241.61.1 Boehringer Ingelheim Investigational Site, Mannheim, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was nonrandomised, open-label and fixed-sequence and was performed in 2 separate groups of 2 periods each in healthy male and female volunteers. Treatments for the two periods were in group 1 cyclosporine (cyclo) and cyclo and faldaprevir (FDV), and in Group 2 tacrolimus (tac) and tac and FDV.
Groups:
- Cyclosporine / Cyclosporine + Faldaprevir: fixed sequence group 1: single dose of 50 mg cyclo on Day 1 in period 1; treated with FDV 240 mg on Day -7 (loading dose) and 120 mg FDV on Days -6 to 7 and a single dose of 50 mg cyclo on Day 1 in period 2. Mode of administration: oral, with 240 mL water after a meal. A washout period of at least 14 days separated administration of cyclo in the treatment periods.
- Tacrolimus / Tacrolimus + Faldaprevir: fixed sequence group 2: single dose of 0.5 mg tac on Day 1 in period 1; treated with FDV 240 mg on Day -7 (loading dose) and 120 mg FDV on Days -6 to 7 and a single dose of 0.5 mg tac on Day 1 in period 2. Mode of administration: oral, with 240 mL water after a meal. A washout period of at least 14 days separated administration of cyclo in the treatment periods.
Period: Cyclo or Tac (Single Dose, Day 1)
Arm/Group | Cyclosporine / Cyclosporine + Faldaprevir | Tacrolimus / Tacrolimus + Faldaprevir
Started | 16 | 16
Completed | 16 | 15
Not Completed | 0 | 1
Not completed — not treated | 0 | 1
Period: Cyclo or Tac (Day 1) + FDV (Day -7 to 7)
Arm/Group | Cyclosporine / Cyclosporine + Faldaprevir | Tacrolimus / Tacrolimus + Faldaprevir
Started | 16 | 15
Completed | 13 | 15
Not Completed | 3 | 0
Not completed — Adverse Event | 1 | 0
Not completed — not specified above | 2 | 0

BASELINE CHARACTERISTICS:
Population: treated set (TS): included all subjects who took at least one dose of study medication during the treatment period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cyclosporine / Cyclosporine + Faldaprevir | Tacrolimus / Tacrolimus + Faldaprevir | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.2 (8.3) | 41.5 (8.8) | 41.3 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: AUC 0-infinity (Area Under the Concentration-time Curve of the Cyclo in Plasma Over the Time Interval From 0 Extrapolated to Infinity)
Description: AUC 0-infinity (area under the concentration-time curve of the cyclo in plasma over the time interval from 0 extrapolated to infinity).
  PK sampling (relative to the first cyclo administration [h:min])
  Period 1:
  for cyclo 0:00h, 0:30h, 1:00h, 1:30h, 2:00h, 3:00h, 4:00h, 6:00h, 8:00h, 10:00h, 12:00h, 16:00h, 24:00h, 48:00h, 72:00h, 96:00h.
  period 2 for cyclo 0:00h, 0:30h, 1:00h, 1:30h, 2:00h, 3:00h, 4:00h, 6:00h, 8:00h, 10:00h, 12:00h, 16:00h, 24:00h, 48:00h, 72:00h, 96:00h, 120:00h, 144:00h, 168:00h.
Time Frame: up to 168 hours (details in description)
Population: pharmacokinetic set of cyclo (PKS cyclo): The subject set for the evaluation of PK endpoints was to include all treated subjects who provided at least 1 observation of cyclo in plasma for at least 1 primary endpoint, and who did not have important protocol violations with respect to the statistical evaluation of PK endpoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Cyclosporine: fixed sequence group 1: treated with cyclo 50 mg on Day 1 in period 1.
- Cyclosporine + Faldaprevir: fixed sequence group 1: treated with FDV 240 mg on Day -7 and 120 mg FDV on Days -6 to 7; single dose of 50 mg cyclo on Day 1 in period 2.
Arm/Group | Cyclosporine | Cyclosporine + Faldaprevir
Number analyzed (Participants) | 16 | 13
ng*h/mL | 672 (17.4) | 732 (25.1)
Statistical Analysis 1: Comparison: Cyclosporine vs Cyclosporine + Faldaprevir; Geometric mean (gMean) ratio of cyclo + FDV to cyclo treatment. The statistical model used for the analysis of primary endpoints was an analysis of variance (ANOVA) model on the logarithmic scale. This model accounted for variation from 'subject' and 'treatment' effects. The 'subject' effect was considered to be random, whereas the 'treatment' effect was considered as fixed; Test type: Non-Inferiority or Equivalence — Null hypothesis (H0): ratio is outside of interval (80%, 125%) vs. alternative hypothesis (H1): ratio is inside of interval (80%, 125%); p = 0.0033, ANOVA; gMean ratio (%) = 108.20, 90% CI 2-sided [99.992 to 117.076], Standard Error of Mean 11.5 — ratio of cyclo + FDV to cyclo treatment. The standard error of the mean actually is the geometric coefficient of variation (%)

2. Primary Outcome: AUC 0-tz (Area Under the Concentration-time Curve of the Cyclo in Plasma Over the Time Interval From 0 to the Last Quantifiable Point)
Description: AUC 0-tz (area under the concentration-time curve of the cyclo in plasma over the time interval from 0 to the last quantifiable point).
  PK sampling (relative to the first cyclo administration [h:min]):
  Period 1:
  for cyclo 0:00h, 0:30h, 1:00h, 1:30h, 2:00h, 3:00h, 4:00h, 6:00h, 8:00h, 10:00h, 12:00h, 16:00h, 24:00h, 48:00h, 72:00h, 96:00h period 2 for cyclo 0:00h, 0:30h, 1:00h, 1:30h, 2:00h, 3:00h, 4:00h, 6:00h, 8:00h, 10:00h, 12:00h, 16:00h, 24:00h, 48:00h, 72:00h, 96:00h, 120:00h, 144:00h, 168:00h.
Time Frame: up to 168 hours (details in description)
Population: PKS cyclo
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Cyclosporine | Cyclosporine + Faldaprevir
Number analyzed (Participants) | 16 | 13
ng*h/mL | 635 (16.2) | 685 (25.2)
Statistical Analysis 1: Comparison: Cyclosporine vs Cyclosporine + Faldaprevir; gMean ratio of cyclo+FDV to cyclo treatment The statistical model used for the analysis of primary endpoints was an analysis of variance (ANOVA) model on the logarithmic scale. This model accounted for variation from 'subject' and 'treatment' effects. The 'subject' effect was considered to be random, whereas the 'treatment' effect was considered as fixed; Test type: Non-Inferiority or Equivalence — H0: ratio is outside of interval (80%, 125%) vs. H1: ratio is inside of interval (80%, 125%); p = 0.0019, ANOVA; gMean ratio (%) = 106.60, 90% CI 2-sided [98.360 to 115.534], Standard Error of Mean 11.7 — gMean ratio of cyclo+FDV to cyclo treatment. The standard error of the mean actually is the geometric coefficient of variation (%)

3. Primary Outcome: Cmax (Maximum Measured Concentration of the Cyclo in Plasma)
Description: Cmax (maximum measured concentration of the cyclo in plasma).
  PK sampling (relative to the first cyclo administration [h:min]):
  Period 1: for cyclo 0:00h, 0:30h, 1:00h, 1:30h, 2:00h, 3:00h, 4:00h, 6:00h, 8:00h, 10:00h, 12:00h, 16:00h, 24:00h, 48:00h, 72:00h, 96:00h period 2 for cyclo 0:00h, 0:30h, 1:00h, 1:30h, 2:00h, 3:00h, 4:00h, 6:00h, 8:00h, 10:00h, 12:00h, 16:00h, 24:00h, 48:00h, 72:00h, 96:00h, 120:00h, 144:00h, 168:00h
Time Frame: up to 168 hours (details in description)
Population: PKS cyclo
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cyclosporine | Cyclosporine + Faldaprevir
Number analyzed (Participants) | 16 | 13
ng/mL | 172 (34.7) | 164 (27.8)
Statistical Analysis 1: Comparison: Cyclosporine vs Cyclosporine + Faldaprevir; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — H0: ratio is outside of interval (80%, 125%) VS H1: ratio is inside of interval (80%, 125%); p = 0.0457, ANOVA; gMean ratio (%) = 90.14, 90% CI 2-sided [80.281 to 101.205], Standard Error of Mean 16.6 — [estimate comment as in outcome 2, analysis 1]

4. Primary Outcome: Cmax,ss (Maximum Measured Concentration of the FDV [Followed by Cyclo Treatment] in Plasma at Steady State Over a Uniform Dosing Interval τ)
Description: Cmax,ss (maximum measured concentration of the FDV [followed by cyclo treatment] in plasma at steady state over a uniform dosing interval τ).
  PK sampling (relative to the first cyclo administration [h:min]):
  period 2 For FDV
  -144:00h, -120:00h, -96:00h, -72:00h, -48:00h, -24:00h, -23:30h, -23:00h, -22:30h, -22:00h, -21:00h, -20:00h, -18:00h, -16:00h, -14:00h, -12:00h, -8:00h, 0:00h, 0:30h, 1:00h, 1:30h, 2:00h, 3:00h, 4:00h, 6:00h, 8:00h, 10:00h, 12:00h, 16:00h, 24:00h, 48:00h, 72:00h, 96:00h, 120:00h, 144:00h, 168:00h
Time Frame: up to 168 hours (details in description)
Population: PKS cyclo + treated with FDV alone (arm: Faldaprevir) or started combination treatment FDV+cyclosporine in treatment period 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Faldaprevir: fixed sequence group 1: treated with FDV 240 mg on Day -7 and 120 mg FDV on Days -6 to 1 [followed by cyclo treatment] in period 2
Arm/Group | Faldaprevir | Cyclosporine + Faldaprevir
Number analyzed (Participants) | 15 | 14
ng/mL | 1740 (225) | 2470 (331)
Statistical Analysis 1: Comparison: Faldaprevir vs Cyclosporine + Faldaprevir; gMean ratio of cyclo+FDV to FDV treatment. The statistical model used for the analysis of primary endpoints was an analysis of variance (ANOVA) model on the logarithmic scale. This model accounted for variation from 'subject' and 'treatment' effects. The 'subject' effect was considered to be random, whereas the 'treatment' effect was considered as fixed; Test type: Non-Inferiority or Equivalence — H0: ratio is outside of interval (80%, 125%) VS H1: ratio is inside of interval (80%, 125%); p = 0.8122, ANOVA; gMean ratio (%) = 140.98, 90% CI 2-sided [111.772 to 177.833], Standard Error of Mean 35.8 — gMean ratio of cyclo+FDV to FDV treatment. The standard error of the mean actually is the geometric coefficient of variation (%)

5. Primary Outcome: C24,ss (Maximum Measured Concentration of the FDV in Plasma at Steady State Over a 24 Hour Dosing Interval)
Description: PK sampling (relative to the first cyclo administration [h:min]):
  period 2 For FDV
  -144:00h, -120:00h, -96:00h, -72:00h, -48:00h, -24:00h, -23:30h, -23:00h, -22:30h, -22:00h, -21:00h, -20:00h, -18:00h, -16:00h, -14:00h, -12:00h, -8:00h, 0:00h, 0:30h, 1:00h, 1:30h, 2:00h, 3:00h, 4:00h, 6:00h, 8:00h, 10:00h, 12:00h, 16:00h, 24:00h, 48:00h, 72:00h, 96:00h, 120:00h, 144:00h, 168:00h
Time Frame: up to 168 hours (details in description)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Faldaprevir | Cyclosporine + Faldaprevir
Number analyzed (Participants) | 15 | 14
ng/mL | 619 (194) | 723 (205)
Statistical Analysis 1: Comparison: Faldaprevir vs Cyclosporine + Faldaprevir; [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority or Equivalence — H0: ratio is outside of interval (80%, 125%) VS H1: ratio is inside of interval (80%, 125%); p = 0.0650, ANOVA; gMean ratio (%) = 116.92, 90% CI 2-sided [108.674 to 125.801], Standard Error of Mean 11.0 — [estimate comment as in outcome 4, analysis 1]

6. Primary Outcome: AUC τ,ss (Area Under the Concentration-time Curve of the Analyte in Plasma at Steady State Over a Uniform Dosing Interval τ)
Description: AUC τ,ss (area under the concentration-time curve of the FDV in plasma at steady state over a uniform dosing interval τ).
  PK sampling (relative to the first cyclo administration [h:min]):
  period 2 For FDV
  -144:00h, -120:00h, -96:00h, -72:00h, -48:00h, -24:00h, -23:30h, -23:00h, -22:30h, -22:00h, -21:00h, -20:00h, -18:00h, -16:00h, -14:00h, -12:00h, -8:00h, 0:00h, 0:30h, 1:00h, 1:30h, 2:00h, 3:00h, 4:00h, 6:00h, 8:00h, 10:00h, 12:00h, 16:00h, 24:00h, 48:00h, 72:00h, 96:00h, 120:00h, 144:00h, 168:00h
Time Frame: up to 168 hours (details in description)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Faldaprevir | Cyclosporine + Faldaprevir
Number analyzed (Participants) | 15 | 14
ng*h/mL | 24600 (196) | 30600 (267)
Statistical Analysis 1: Comparison: Faldaprevir vs Cyclosporine + Faldaprevir; [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority or Equivalence — H0: ratio is outside of interval (80%, 125%) VS H1: ratio is inside of interval (80%, 125%); p = 0.4181, ANOVA; gMean ratio (%) = 122.68, 90% CI 2-sided [104.80 to 143.60], Standard Error of Mean 23.9 — [estimate comment as in outcome 4, analysis 1]

7. Primary Outcome: AUC 0-infinity (Area Under the Concentration-time Curve of the Tac in Plasma Over the Time Interval From 0 Extrapolated to Infinity)
Description: AUC 0-infinity (area under the concentration-time curve of the tac in plasma over the time interval from 0 extrapolated to infinity).
  PK sampling (relative to the first tac administration):
  Period 1: for tac 0:00h, 0:30h, 1:00h, 1:30h, 2:00h, 3:00h, 4:00h, 6:00h, 8:00h, 10:00h, 12:00h, 16:00h, 24:00h, 48:00h, 72:00h, 96:00h, 144:00h, 168:00h, 192:00h period 2 for tac
  -192:00h, -168:00h, 0:00h, 0:30h, 1:00h, 1:30h, 2:00h, 3:00h, 4:00h, 6:00h, 8:00h, 10:00h, 12:00h, 16:00h, 24:00h, 48:00h, 72:00h, 96:00h, 120:00h, 144:00h, 168:00h
Time Frame: up to 192 hours (details in description)
Population: pharmacokinetic set of tac (PKS tac): The subject set for the evaluation of PK endpoints was to include all treated subjects who provided at least 1 observation of tac in plasma for at least 1 primary endpoint, and who did not have important protocol violations with respect to the statistical evaluation of PK endpoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Tacrolimus: fixed sequence group 2: treated with tac 0.5 mg on Day 1 in period 1.
- Tacrolimus + Faldaprevir: fixed sequence group 2: treated with FDV 240 mg on Day -7 and 120 mg FDV on Days -6 to 7; single dose of 0.5 mg tac on Day 1 in period 2.
Arm/Group | Tacrolimus | Tacrolimus + Faldaprevir
Number analyzed (Participants) | 15 | 15
ng*h/mL | 16.0 (57.6) | 20.4 (62.9)
Statistical Analysis 1: Comparison: Tacrolimus vs Tacrolimus + Faldaprevir; gMean ratio of tac+FDV to FDV treatment. The statistical model used for the analysis of primary endpoints was an analysis of variance (ANOVA) model on the logarithmic scale. This model accounted for variation from 'subject' and 'treatment' effects. The 'subject' effect was considered to be random, whereas the 'treatment' effect was considered as fixed; Test type: Non-Inferiority or Equivalence — H0: ratio is outside of interval (80%, 125%) VS H1: ratio is inside of interval (80%, 125%); p = 0.6207, ANOVA; gMean ratio (%) = 127.41, 90% CI 2-sided [114.453 to 141.827], Standard Error of Mean 16.8 — gMean ratio of tac+FDV to FDV treatment. The standard error of the mean actually is the geometric coefficient of variation (%)

8. Primary Outcome: AUC 0-tz (Area Under the Concentration-time Curve of the Tac in Plasma Over the Time Interval From 0 to the Last Quantifiable Point)
Description: AUC 0-tz (area under the concentration-time curve of the tac in plasma over the time interval from 0 to the last quantifiable point).
  PK sampling (relative to the first tac administration [h:min]):
  Period 1: for tac
  0:00h, 0:30h, 1:00h, 1:30h, 2:00h, 3:00h, 4:00h, 6:00h, 8:00h, 10:00h, 12:00h, 16:00h, 24:00h, 48:00h, 72:00h, 96:00h, 144:00h, 168:00h, 192:00h
  Period 2 For tac
  -192:00h, -168:00h, 0:00h, 0:30h, 1:00h, 1:30h, 2:00h, 3:00h, 4:00h, 6:00h, 8:00h, 10:00h, 12:00h, 16:00h, 24:00h, 48:00h, 72:00h, 96:00h, 120:00h, 144:00h, 168:00h
Time Frame: up to 192 hours (details in description)
Population: PKS tac
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Tacrolimus | Tacrolimus + Faldaprevir
Number analyzed (Participants) | 15 | 15
ng*h/mL | 11.1 (62.8) | 15.3 (66.2)
Statistical Analysis 1: Comparison: Tacrolimus vs Tacrolimus + Faldaprevir; [analysis description as in outcome 7, analysis 1]; Test type: Non-Inferiority or Equivalence — H0: ratio is outside of interval (80%, 125%) VS H1: ratio is inside of interval (80%, 125%); p = 0.8592, ANOVA; gMean ratio (%) = 136.85, 90% CI 2-sided [118.683 to 157.793], Standard Error of Mean 22.4 — [estimate comment as in outcome 7, analysis 1]

9. Primary Outcome: Cmax (Maximum Measured Concentration of the Tac in Plasma)
Description: Cmax (maximum measured concentration of the tac in plasma).
  PK sampling (relative to the first tac administration [h:min]):
  Period 1:
  for tac 0:00h, 0:30h, 1:00h, 1:30h, 2:00h, 3:00h, 4:00h, 6:00h, 8:00h, 10:00h, 12:00h, 16:00h, 24:00h, 48:00h, 72:00h, 96:00h, 144:00h, 168:00h, 192:00h Period 2 For tac
  -192:00h, -168:00h, 0:00h, 0:30h, 1:00h, 1:30h, 2:00h, 3:00h, 4:00h, 6:00h, 8:00h, 10:00h, 12:00h, 16:00h, 24:00h, 48:00h, 72:00h, 96:00h, 120:00h, 144:00h, 168:00h
Time Frame: up to 192 hours (details in description)
Population: PKS tac
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Tacrolimus + Faldaprevir: fixed sequence group 2: treated with tac 0.5 mg on Day 1 in period 1, treated with FDV 240 mg on Day -7 and 120 mg FDV on Days -6 to 7; single dose of 0.5 mg tac on Day 1 in period 2.
Arm/Group | Tacrolimus | Tacrolimus + Faldaprevir
Number analyzed (Participants) | 15 | 15
ng/mL | 1.14 (35.5) | 1.13 (48.9)
Statistical Analysis 1: Comparison: Tacrolimus vs Tacrolimus + Faldaprevir; [analysis description as in outcome 7, analysis 1]; Test type: Non-Inferiority or Equivalence — H0: ratio is outside of interval (80%, 125%) VS H1: ratio is inside of interval (80%, 125%); p = 0.0269, ANOVA; gMean ratio (%) = 99.15, 90% CI 2-sided [82.857 to 118.644], Standard Error of Mean 28.5 — [estimate comment as in outcome 7, analysis 1]

10. Primary Outcome: Cmax,ss (Maximum Measured Concentration of the FDV [Followed by Tac Treatment] in Plasma at Steady State Over a Uniform Dosing Interval τ)
Description: Cmax,ss (maximum measured concentration of the FDV [followed by tac treatment] in plasma at steady state over a uniform dosing interval τ).
  PK sampling (relative to the first tac administration [h:min]):
  period 2 For FDV
  -144:00h, -120:00h, -96:00h, -72:00h, -48:00h, -24:00h, -23:30h, -23:00h, -22:30h, -22:00h, -21:00h, -20:00h, -18:00h, -16:00h, -14:00h, -12:00h, -8:00h, 0:00h, 0:30h, 1:00h, 1:30h, 2:00h, 3:00h, 4:00h, 6:00h, 8:00h, 10:00h, 12:00h, 16:00h, 24:00h, 48:00h, 72:00h, 96:00h, 120:00h, 144:00h, 168:00h.
Time Frame: up to 168 hours (details in description)
Population: PKS tac
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Faldaprevir: fixed sequence group 2: treated with FDV 240 mg on Day -7 and 120 mg FDV on Days -6 to 1 [followed by tac treatment] in period 2
Arm/Group | Faldaprevir | Tacrolimus + Faldaprevir
Number analyzed (Participants) | 15 | 15
ng/mL | 3120 (35.7) | 2930 (51.3)
Statistical Analysis 1: Comparison: Faldaprevir vs Tacrolimus + Faldaprevir; [analysis description as in outcome 7, analysis 1]; Test type: Non-Inferiority or Equivalence — H0: ratio is outside of interval (80%, 125%) VS H1: ratio is inside of interval (80%, 125%); p = 0.0493, ANOVA; gMean ratio (%) = 93.85, 90% CI 2-sided [80.059 to 110.022], Standard Error of Mean 25.1 — [estimate comment as in outcome 7, analysis 1]

11. Primary Outcome: C24,ss (Maximum Measured Concentration of the FDV [Followed by Tac Treatment] in Plasma at Steady State Over a 24 Hour Dosing Interval)
Description: PK sampling (relative to the first tac administration [h:min]):
  period 2 For FDV
  -144:00h, -120:00h, -96:00h, -72:00h, -48:00h, -24:00h, -23:30h, -23:00h, -22:30h, -22:00h, -21:00h, -20:00h, -18:00h, -16:00h, -14:00h, -12:00h, -8:00h, 0:00h, 0:30h, 1:00h, 1:30h, 2:00h, 3:00h, 4:00h, 6:00h, 8:00h, 10:00h, 12:00h, 16:00h, 24:00h, 48:00h, 72:00h, 96:00h, 120:00h, 144:00h, 168:00h.
Time Frame: up to 168 hours (details in description)
Population: PKS tac
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Faldaprevir: fixed sequence group 2: treated with FDV 240 mg on Day -7 and 120 mg FDV on Days -6 to 7 [followed by tac treatment] in period 2.
Arm/Group | Faldaprevir | Tacrolimus + Faldaprevir
Number analyzed (Participants) | 15 | 15
ng/mL | 904 (56.1) | 900 (52.1)
Statistical Analysis 1: Comparison: Faldaprevir vs Tacrolimus + Faldaprevir; [analysis description as in outcome 7, analysis 1]; Test type: Non-Inferiority or Equivalence — H0: ratio is outside of interval (80%, 125%) VS H1: ratio is inside of interval (80%, 125%); p = 0.0000, ANOVA; gMean ratio (%) = 99.54, 90% CI 2-sided [93.375 to 106.115], Standard Error of Mean 10.0 — [estimate comment as in outcome 7, analysis 1]

12. Primary Outcome: AUC τ,ss (Area Under the Concentration-time Curve of the FDV [Followed by Tac Treatment] in Plasma at Steady State Over a Uniform Dosing Interval τ)
Description: AUC τ,ss (area under the concentration-time curve of the FDV [followed by tac treatment] in plasma at steady state over a uniform dosing interval τ).
  PK sampling (relative to the first cyclo administration [h:min]):
  period 2 For FDV
  -144:00h, -120:00h, -96:00h, -72:00h, -48:00h, -24:00h, -23:30h, -23:00h, -22:30h, -22:00h, -21:00h, -20:00h, -18:00h, -16:00h, -14:00h, -12:00h, -8:00h, 0:00h, 0:30h, 1:00h, 1:30h, 2:00h, 3:00h, 4:00h, 6:00h, 8:00h, 10:00h, 12:00h, 16:00h, 24:00h, 48:00h, 72:00h, 96:00h, 120:00h, 144:00h, 168:00h.
Time Frame: up to 168 hours (details in description)
Population: PKS tac
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Faldaprevir | Tacrolimus + Faldaprevir
Number analyzed (Participants) | 15 | 15
ng*h/mL | 40300 (39.1) | 38700 (48.3)
Statistical Analysis 1: Comparison: Faldaprevir vs Tacrolimus + Faldaprevir; [analysis description as in outcome 7, analysis 1]; Test type: Non-Inferiority or Equivalence — H0: ratio is outside of interval (80%, 125%) VS H1: ratio is inside of interval (80%, 125%); p = 0.0008, ANOVA; gMean ratio (%) = 96.16, 90% CI 2-sided [88.53 to 104.45], Standard Error of Mean 12.9 — [estimate comment as in outcome 7, analysis 1]

ADVERSE EVENTS:
Time Frame: from the date of start trial medication to 28 days after the last trial medication.
Description: Group 1: 16 subjects (sub) treated with cyclosporine (cyclo). After a washout phase the second period started. 15 sub. treated with Faldaprevir (FDV) (Day -7 to 7); 14 subjects treated with a cyclo on Day 1. Group 2: 15 of 16 sub. treated with tacrolimus (tac). After the washout in the second period 15 sub. were treated with FDV alone and FDV+tac.
Groups:
- Cyclosporine (Cyclo): Cyclosporine (cyclo) 50 mg
- Tacrolimus (Tac): Tacrolimus (tac) 0.5 mg
- FDV (ff Cyclo): FDV 120 mg (followed by cyclosporine)
- FDV (ff Tac): FDV 120 mg (followed by tacrolimus)
- Cyclo+FDV: Cyclosporine 50 mg + FDV 120 mg
- Tac+FDV: Tacrolimus 0.5 mg + FDV 120 mg
Arm/Group | Cyclosporine (Cyclo) | Tacrolimus (Tac) | FDV (ff Cyclo) | FDV (ff Tac) | Cyclo+FDV | Tac+FDV
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15 | 0/15 | 0/15 | 0/14 | 1/15
Other Adverse Events (participants affected / at risk) | 6/16 | 5/15 | 10/15 | 7/15 | 4/14 | 5/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cyclosporine (Cyclo) (N=16) | Tacrolimus (Tac) (N=15) | FDV (ff Cyclo) (N=15) | FDV (ff Tac) (N=15) | Cyclo+FDV (N=14) | Tac+FDV (N=15)
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cyclosporine (Cyclo) (N=16) | Tacrolimus (Tac) (N=15) | FDV (ff Cyclo) (N=15) | FDV (ff Tac) (N=15) | Cyclo+FDV (N=14) | Tac+FDV (N=15)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ocular icterus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 2
Eye pruritus (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 2 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 3 | 3 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 1 | 0
Feeling hot (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rash pustular (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Incorrect dose administered (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 5 | 3 | 3 | 4 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are NOT employed by the organization sponsoring the study. There IS an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed.